CLINICAL TRIAL: NCT02031094
Title: The Effect of Liver Regeneration on Resting Energy Expenditure After Liver Resectional Surgery
Brief Title: Energy Expenditure and Regeneration Following Liver Resection Resection
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Royal College of Surgeons of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 13/SS/0019; 2013/R/END/01 (Other: NHS Lothian)
Record Dates: First submitted 2013-11-21; First posted 2014-01-09 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Liver Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major resection: Patients undergoing resection of >3 segments (resting energy expenditure measured by Sense Wear Armband and indirect calorimetry)
  Interventions: Other: Observational study: Sense Wear armband and indirect calorimetry used to measure resting energy expenditure
- Minor resection: Patients undergoing resection of </= 3 segments (resting energy expenditure measured by Sense Wear Armband and indirect calorimetry)
  Interventions: Other: Observational study: Sense Wear armband and indirect calorimetry used to measure resting energy expenditure

INTERVENTIONS:
Other: Observational study: Sense Wear armband and indirect calorimetry used to measure resting energy expenditure — Observational methods of measuring resting energy expenditure

SUMMARY:
This observational study will measure resting energy expenditure in patients who have undergone liver resection and compare methods of measuring resting energy expenditure.

DETAILED DESCRIPTION:
Penetrating liver injury occurs commonly in victims of battlefield trauma. It is associated with a high mortality and morbidity rate. Management of liver injury is complex and challenging and can often involve debridement or anatomical resection of liver tissue.

Following liver resection, the liver regenerates to its original volume. Liver regeneration involves complex metabolic processes and maximal regeneration occurs over the first post operative week. This process is highly energy dependent and adds a further burden on post operative energy and therefore nutritional requirements.

Inadequate post-operative nutrition is associated with poorer outcomes and complication rates. Additionally, over feeding is also associated with adverse outcome. The actual additional energy expenditure involved in liver regeneration is not currently known and therefore accurate calorific balance remains a challenge.

The measurement of energy expenditure in these patients is therefore important. Traditionally energy expenditure has been measured by indirect calorimetry and doubly labelled water. These techniques require skilled operators and are often impractical for everyday clinical usage and impossible in the deployed setting.

A recent development is a lightweight armband that measures total and resting energy expenditure. It has been validated against the gold standard techniques in various settings including cancer cachexia, obesity and healthy volunteers and is deemed highly acceptable also. It has not been validated in the unique setting of liver regeneration.

Therefore this study will assess the energy expenditure in patients undergoing liver regeneration and attempt to validate a new minimally invasive device against the traditional measurements of energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing liver resection for benign or malignant hepatic neoplasm

Exclusion Criteria:

* Inability to give written, informed consent.
* Jaundice (Bilirubin > 100 μmol/L)
* Liver resection combined with secondary surgical procedure.
* Age < 18 years
* Pregnant women
* Unable to tolerate either measuring device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hepatic resection for benign or malignant neoplasms.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Resting Energy Expenditure (Kcal) following liver resection | 2 weeks pre-operatively and post-operative days 3,5 and 7

SECONDARY OUTCOMES:
Change in total energy expenditure (Kcal) following liver resection | 2 weeks pre-operatively and post-operative days 3,5 and 7

OTHER OUTCOMES:
Volume of liver resected (g) | Post operative day 1
Resting energy expenditure (REE) (Kcal) | 4 weeks post-operative
Post-operative blood tests (FBC, U&E, LFT, Coag) | Post-operative days 1-7
Complications | Day of surgery and post-operative days 1-30

CONTACTS AND LOCATIONS:
Overall Officials: Michael j Hughes, Principal Investigator — University of Edinburgh; Stephen J Wigmore, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom